CLINICAL TRIAL: NCT00005803
Title: A Phase I/II Study of Autologous Stem Cell Transplantation Followed by Nonmyeloablative Allogeneic Stem Cell Transplantation for Patients With Relapsed or Refractory Lymphoma - A Multi-center Trial
Brief Title: Autologous Stem Cell Transplant Followed by Donor Stem Cell Transplant in Treating Patients With Relapsed or Refractory Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1409.00; NCI-2010-00130 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1409.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2000-06-02; First posted 2003-01-27 (Estimated); Results first posted 2017-12-07 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2019-12

CONDITIONS: Prolymphocytic Leukemia; Recurrent Adult Hodgkin Lymphoma; Recurrent Childhood Hodgkin Lymphoma; Recurrent Childhood Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Non-Hodgkin Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; Refractory Small Lymphocytic Lymphoma; T-Cell Chronic Lymphocytic Leukemia; T-Cell Prolymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Leukemia, Prolymphocytic, T-Cell | interventions — Carmustine; carmustine, poliferprosan 20 drug combination; Cyclophosphamide; Cyclosporine; Cyclosporins; Cytarabine; Etoposide; fludarabine phosphate; Melphalan; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (tandem transplantation) (Experimental): See Detailed Description
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Procedure: Autologous-Allogeneic Tandem Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cyclophosphamide; Drug: Cyclosporine; Drug: Cytarabine; Drug: Etoposide; Drug: Fludarabine Phosphate; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Biological: Therapeutic Autologous Lymphocytes; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous transplantation
  Other Names: Autologous Stem Cell Transplantation
Procedure: Autologous-Allogeneic Tandem Hematopoietic Stem Cell Transplantation — Undergo autologous-allogeneic tandem hematopoietic stem cell transplantation
  Other Names: auto-allo HCT
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; Oforta; SH T 586
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic transplantation
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Biological: Therapeutic Autologous Lymphocytes — IV donor lymphocyte infusion
  Other Names: Autologous T-cells
Radiation: Total-Body Irradiation — Undergo radiotherapy
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase I/II trial studies how well autologous stem cell transplant followed by donor stem cell transplant works in treating patients with lymphoma that has returned or does not respond to treatment. Peripheral blood stem cell transplant using stem cells from the patient or a donor may be able to replace immune cells that were destroyed by chemotherapy used to kill cancer cells. The donated stem cells may also help destroy any remaining cancer cells (graft-versus-tumor effect).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate engraftment of human leukocyte antibody (HLA) identical peripheral blood stem cell (PBSC) allografts given after conditioning with total-body irradiation (TBI) (200cGy) +/- fludarabine (fludarabine phosphate), 90 mg/m^2 and post-grafting immunosuppression with cyclosporine (CSP)/mycophenolate mofetil (MMF) in refractory or relapsed lymphoma patients following an initial autologous peripheral blood stem cell transplant (PBSCT) for disease cytoreduction.

II. To determine the non-relapse mortality at day 100 post-non-myeloablative allografting following mobilization and high-dose chemotherapy with autografting.

SECONDARY OBJECTIVES:

I. To determine the disease free survival and overall survival of non-myeloablative allografting following autologous PBSCT.

OUTLINE:

CONDITIONING REGIMEN: Patients with matched, related stem cell donors receive cyclophosphamide intravenously (IV) on days -6 and -5 and undergo TBI twice daily (BID) on days -3 to -1. Patients with matched, unrelated stem cell donors receive carmustine IV over 3 hours on day -7, etoposide IV over 2 hours BID on days -6 to -3, and cytarabine IV over 3 hours BID on days -6 to -3, and melphalan IV over 30 minutes on day -2.

TRANSPLANTATION: All patients undergo autologous PBSCT on day 0.

NON-MYELOABLATIVE CONDITIONING: Beginning 40-120 days following PBSC transplant, patients with related donors undergo TBI on day 0. Patients with unrelated donors receive fludarabine phosphate IV over 30 minutes on days -4 to -2 and undergo TBI on day 0.

TRANSPLANTATION: Patients undergo non-myeloablative allogeneic PBSCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) BID on days -3 to 56 (patients with related donors) or 100 (patients with unrelated donors) followed by taper to day 180. Patients also receive mycophenolate mofetil PO BID on days 0-27 (patients with related donors) or thrice daily (TID) on days 0-27, then BID on days 28-40 followed by taper to day 96 (patients with unrelated donors).

Some patients may undergo donor lymphocyte infusion if there is evidence of disease progression and no evidence of graft-vs-host disease (GVHD).

After completion of study treatment, patients are followed up at day 180, 1 year, 1.5 years, 2 years, 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients with lymphoma (non-Hodgkin lymphoma [NHL], chronic lymphocytic leukemia/small lymphocytic lymphoma [CLL/SLL] or Hodgkin's lymphoma) with primary refractory or relapsed disease after standard chemotherapy at high risk of relapse with conventional autografting; patients with a diagnosis of CLL (or small lymphocytic lymphoma) or diagnosis of CLL that progresses to prolymphocytic leukemia (PLL), or T-cell CLL or PLL
* Must have an HLA genotypically or phenotypically identical related donor or, at a minimum, a high likelihood of identifying an HLA-matched unrelated donor; the determination of availability of a suitable unrelated donor may be based on a World-Book search
* Cross-over to other tandem autologous-allogeneic research protocol (#2241) will be allowed if the patient loses the suitable HLA-matched related or unrelated donor but has an available HLA-haploidentical donor before receiving the allogeneic transplantation and if the patient meets the eligibility criteria of the subsequent study
* Cross-over from other tandem autologous-allogeneic research protocol (#2241) will be allowed if a suitable HLA-matched related or unrelated donor is identified before receiving the allogeneic transplantation and if the patient meets the eligibility criteria of the subsequent study
* Signed informed consent
* Detectable tumor on radiographic studies or bone marrow biopsy prior to mobilization regimen
* Expected survival >= 3 months from study entry
* DONOR: HLA genotypically or phenotypically identical related donor
* DONOR: Must consent to granulocyte-colony stimulating factor (G-CSF) (filgrastim) administration and leukapheresis for both PBSC allograft and subsequent donor lymphocyte infusion (DLI)
* DONOR: Must have adequate veins for leukapheresis or agree to placement of central venous catheter (femoral or subclavian)
* DONOR: Age < 75 years (yrs), older donors may be considered after review at Patient Care Conference
* DONOR: Fred Hutchinson Cancer Research Center (FHCRC) matching allowed will be grades 1.0 to 2.1; unrelated donors who are prospectively: matched for HLA-A, B, C, DRB1 and DQB1 by high resolution typing; only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: Donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before HCT; if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results; a positive anti-donor cytotoxic crossmatch is an absolute donor exclusion
* DONOR: Patient and donor pairs homozygous at a mismatched allele in the graft rejection vector are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* DONOR: Only G-CSF mobilized peripheral blood mononuclear cells (PBMC) only will be permitted as a hematopoietic stem cell (HSC) source on this protocol

Exclusion Criteria:

* Life expectancy severely limited by disease other than lymphoma
* Prior autologous hematopoietic stem cell transplant
* Patients at high risk of veno-occlusive disease of the liver (criteria not yet rigorously defined but includes bilirubin > 2.0 mg and serum glutamic oxaloacetic transaminase [SGOT] or serum glutamate pyruvate transaminase [SGPT] > 2 x normal); patients may be accepted outside of this range if cleared by gastrointestinal (GI) consult
* Cardiac ejection fraction (EF) < 40% on multi-gated acquisition (MUGA) scan or cardiac echocardiogram (echo) (or if unable to obtain ejection fraction, shortening fraction of < 26%); patients with active or a history of cardiac disease should be evaluated with appropriate cardiac studies and/or consult; ejection fraction is required if age > 50 years or there is a history of anthracyclines or history of cardiac disease; patients with a shortening fraction < 26% may be enrolled if approved by a cardiologist
* Baseline serum-creatinine > 2.0 mg/dl and a calculated or measured creatinine clearance of < 50 ml/minute
* Seropositive for the human immunodeficiency virus (HIV)
* Pulmonary dysfunction as measured by a corrected diffusing capacity of the lung for carbon monoxide (DLCO) < 50% of predicted total lung capacity (TLC) < 30%, forced expiratory volume in 1 second (FEV1) < 30% and/or receiving supplementary continuous oxygen; the FHCRC principal investigator (PI) of the study must approve enrollment of all patients with pulmonary nodules
* Pregnancy or breast-feeding
* Patients with poorly controlled hypertension despite hypertensive medication
* Karnofsky score less than 60; pediatric criteria: Lansky Play-Performance Score < 40
* Patients with cluster of differentiation (CD)34 selected auto grafts
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers); this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence; this exclusion does not apply to patients with non-hematologic malignancies that do not require therapy
* DONOR: Identical twin
* DONOR: Age less than 12 years
* DONOR: Pregnancy
* DONOR: Human immunodeficiency virus (HIV) seropositivity
* DONOR: Inability to achieve adequate venous access
* DONOR: Known allergy to G-CSF
* DONOR: Current serious systemic illness
* DONOR: Failure to meet FHCRC criteria for stem cell donation
* DONOR: Donor (or centers) who will exclusively donate marrow

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 1999-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Maloney, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (5):
- United States (4):
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - VA Puget Sound Health Care System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
- Universitaet Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Tandem Transplantation)
Started | 76
Completed | 54
Not Completed | 22

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Tandem Transplantation)
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 75
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 72
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Engraftment of HLA Identical PBSC Allografts
Description: Number of patients who engrafted by Day 56 post allogeneic transplant. Failure to engraft is defined as the absence of detectable donor cells in the marrow. The rates and accompanying confidence intervals associated with failure of engraftment at day +56 will be calculated after every 5th patient is enrolled on the study. If the lower limit to the appropriate one-sided 80% confidence interval exceeds 25%, this will be considered sufficient evidence of an excess "failure" rate and the study will be stopped. For these purposes, all patients will be evaluated together (patients with chemosensitive and chemoresistant disease).
Time Frame: Day 56
Population: Only includes patients who received allo transplant. One patient is excluded because they did not survive long enough to test for engraftment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tandem Transplantation)
Number analyzed (Participants) | 53
Participants | 53

2. Primary Outcome: Non-Relapse Mortality
Description: The rates and accompanying confidence intervals associated with transplant-related mortality will be calculated after every 5th patient is enrolled on the study. If the lower limit to the appropriate one-sided 80% confidence interval exceeds 25%, this will be considered sufficient evidence of an excess "failure" rate and the study will be stopped. For these purposes, all patients will be evaluated together (patients with chemosensitive and chemoresistant disease).
Time Frame: Day 100 post-non-myeloablative allografting following mobilization and high-dose chemotherapy with autografting
Population: Although 54 patients received both auto transplant & allo transplant, one patient did not survive to day 100.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Tandem Transplantation)
Number analyzed (Participants) | 53
Participants | 3

3. Secondary Outcome: Overall Survival (OS)
Description: Number of patients surviving by interval. Chemosensitive and chemoresistant subjects will be analyzed separately.
Time Frame: From the date of autologous transplant until the time of death, assessed up to 3 years
Population: One patient who counted to accrual is not included here. They received conditioning for autologous transplant, but then did not receive the transplant.
Measure: Count of Participants; unit: Participants
Groups:
- Chemosensitive Group: Patients who were CR or PR to most recent chemotherapy regimen.
- Chemoresistant Group: Patients who were not CR or PR to most recent chemotherapy regimen.
- Unknown Chemosensitivity Group: Patients who could not be evaluated for chemosensitivity.
Arm/Group | Chemosensitive Group | Chemoresistant Group | Unknown Chemosensitivity Group
Number analyzed (Participants) | 51 | 22 | 2
Participants
  6 Months | 39 | 14 | 1
  1 Year | 31 | 10 | 0
  1.5 Years | 27 | 9 | 0
  2 Years | 26 | 8 | 0
  3 Years | 23 | 8 | 0

4. Secondary Outcome: Progression Free-survival (PFS)
Description: Number of patients surviving without disease by interval. Chemosensitive and chemoresistant subjects will be analyzed separately.
Time Frame: From the date of autologous transplant until the time of progression, relapse, death, or the date the patient was last known to be in remission, assessed up to 3 years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Chemosensitive Group | Chemoresistant Group | Unknown Chemosensitivity Group
Number analyzed (Participants) | 51 | 22 | 2
Participants
  6 Months | 36 | 12 | 1
  1 Year | 27 | 8 | 0
  1.5 Years | 25 | 8 | 0
  2 Years | 25 | 8 | 0
  3 Years | 22 | 8 | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Tandem Transplantation)
Serious Adverse Events (participants affected / at risk) | 10/76
Other Adverse Events (participants affected / at risk) | 24/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tandem Transplantation) (N=76)
Bowel perforation and sepsis (Infections and infestations) | 1 (1)
Sepsis with respiratory failure and mental status changes (Infections and infestations) | 1 (1)
Tachycardia, intubation, sepsis and pulmonary embolus (Infections and infestations) | 1 (1)
Death due to multiple pulmonary infections (Infections and infestations) | 1 (1)
Pulmonary failure requiring intubation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Death due to infection with pericardial and epicardial involvement (Infections and infestations) | 1 (1)
Respiratory arrest due to disease progression (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia due to organizing pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxemia during PBSC infusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intra-abdominal hemorrhage when undergoing VATS procedure (Surgical and medical procedures) | 1 (1)
Seizures (General disorders) | 1 (1) — no etilogy for the seizures identified
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Tandem Transplantation) (N=76)
Hyperbilirubinemia (Hepatobiliary disorders) | 11 (11)
Increased Creatinine (Renal and urinary disorders) | 16 (16)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (10)
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes